CLINICAL TRIAL: NCT03435822
Title: Clinical Study on Chinese Children's Asthma Action Plan
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Children's Hospital (Other)
Collaborators: Tian Jing Children's Hospital (Unknown); Capital Institute of Pediatrics, China (Other); Peking University Third Hospital (Other); Beijing Tsinghua Chang Gung Hospital (Other); Tianjin Medical University Second Hospital (Other); Peking University Bin Hai Hospital (Unknown); The First Hospital of Qinhuangdao (Other Government); Tangshan Maternal and Child Health Hospital (Other); Children's Hospital of Hebei Province (Other)
Responsible Party: Principal Investigator, Kunling Shen, Chief of China National Clinical Research Center for Respiratory Diseases, Beijing Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCHlung009
Record Dates: First submitted 2018-02-12; First posted 2018-02-19 (Actual); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Asthma in Children
Keywords: asthma; children; action plan; China; CCAAP
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- asthma action plan management group (Other): Patients in this group will be provided both written asthma action plan and mobile-based APP to remind them take medicine regularly and direct them what to do when asthma get worse.
  Interventions: Other: asthma action plan management group
- conventional management group (Other): Patients in this group will be provided conventional management method with prescriptions and asthma diaries.
  Interventions: Other: conventional management group

INTERVENTIONS:
Other: asthma action plan management group — Patients will follow the directions in asthma action plan when their asthma get worse.
  Other Names: conventional management group
  Arms: asthma action plan management group
Other: conventional management group — Patients will follow the directions in conventional strategy when their asthma get worse.
  Arms: conventional management group

SUMMARY:
This study is a multi-center randomized controlled trial of children with asthma. The objective of the study is to assess the efficacy of China Children Asthma Action Plan (CCAAP), which is the first asthma action plan for children with asthma in China, in asthma management.

DETAILED DESCRIPTION:
Asthma is the most common chronic illness of childhood. Asthma action plans have been recommended internationally for more than 20 years by the Global Initiative for Asthma and have been shown to improve asthma-related outcomes. The first asthma action plan for children with asthma in China, which is termed China Children Asthma Action Plan（CCAAP）, as well as a mobile phone-based asthma self management application(APP), were developed recently.

The objective of the study is to assess the efficacy of CCAAP in asthma management.

The study is a multi-center prospective case-controlled study.The enrollment period is 3 months. Patients who is in 6-14 years of age will be randomized recruited into two groups: the asthma action plan group and the conventional group. Patients in asthma action plan group will receive written CCAAP and mobile phone-based asthma self-management APP (Youran Respiratory) which includes an electronic asthma action plan, peak expiratory flow monitor system and Peak Expiratory Flow Meter. Patients in conventional management group will write down the symptoms and PEF in asthma diary. The data of the number of asthma episodes, the improvement of FEV1 , the number of unscheduled medical visits, the score of children's quality of life, the questionnaire of asthma knowledge, ACT / C-ACT score, the absent days of parental work, the absent days of children study, and the cost of health economics will be collected regularly in a year with the interval of 3 months to assess the efficacy of CCAAP in asthma management. The study will recruit 200 cases for each group from ten children's hospitals. The study will be completed in a year.

ELIGIBILITY:
Inclusion Criteria:

* did not receive control treatment or did not reach well-control;
* can perform spirometry pulmonary function tests;
* parents are skilled in using smartphones and APP apps (Android or IOS).

Exclusion Criteria:

* reach the level of asthma control;
* can not use the smartphone APP software;
* can not cooperate the test of peak expiratory flow;
* did not treatment coexist respiratory disease effectively (such as sinusitis, obstructive sleep apnea-hypopnea syndrome, etc.);
* combined with other systemic diseases outside the respiratory system (such as leukemia, rheumatoid arthritis, etc.).
* receiving allergen-specific immunotherapy.
* undergoing trial for other medications or instruments.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2018-03-22 (Estimated); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
number of acute episodes of asthma | 1 year
  number of acute episodes of asthma in a year

SECONDARY OUTCOMES:
the changes of FEV1 before and after management | 1 year
  the changes of FEV1 before and after management in a year
the score of children's quality of life | 1 year
  pediatric asthma quality of life questionnaire contains 23 items in three domains, activity limitation（10）, symptoms（5） and emotional function（8）. The scale from 1-7 for each question. And the higher score the better quality of life.
asthma knowledge | 1 year
  Knowledge, attitude and practice(KAP) questionnaire，contains 27 questions. Multivariate analysis will be carry out based on the answers to questions
ACT / C-ACT score | 1 year
  the change of ACT / C-ACT score. there are 5 questions. For each questions, score ranks from 1 to five. Total score 25: well control, 20~24: control, less than 20: un ncontrol
the absent days of school | 1 year
  the number of absent days of school because of asthma attack
the absent days of parents' work | 1 year
  the number of absent days of parents' work because of children's asthma attack
the cost of health economics | 1 year
  the cost of acute asthma exacerbation in a year
the number of unscheduled medical care | 1 year
  the number of unscheduled medical care in a year

CONTACTS AND LOCATIONS:
Overall Officials: kunling Shen, MD,PhD, Principal Investigator — Beijing Children's Hospital of Capital Medical University

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant available to other researchers so far.